CLINICAL TRIAL: NCT03126682
Title: Effect of Bupropion on Seizure Threshold in Depressed Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00078738
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: MDD
Keywords: Wellbutrin; Electroconvulsive therapy; Right Unilateral Ultra Brief
MeSH Terms: interventions — Bupropion

STUDY DESIGN:
Intervention Model Description: 2 Arms of randomization - one wherein patients get Wellbutrin in first ECT and another arm wherein patients get it with second ECT. Counterbalanced randomization
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Blinding to be done - Outcome assessor and care provider will be blinded to randomization arm of subject
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Wellbutrin during ECT 1 (Active Comparator): Drug - Wellbutrin SR 300Mg Extended-Release Tablet during ECT session 1
  Interventions: Drug: Wellbutrin SR 300Mg Extended-Release Tablet
- Wellbutrin during ECT 2 (Active Comparator): Drug - Wellbutrin SR 300Mg Extended-Release Tablet during ECT session 2.
  Interventions: Drug: Wellbutrin SR 300Mg Extended-Release Tablet

INTERVENTIONS:
Drug: Wellbutrin SR 300Mg Extended-Release Tablet — Wellbutrin SR 300Mg Extended-Release Tablet
  Other Names: Bupropion sustained release formulation

SUMMARY:
The purpose of the study is to examine the effect of bupropion on seizure threshold and duration in depressed patients receiving right unilateral ultra-brief electroconvulsive therapy (ECT). The investigators plan to recruit 10 patients into the study, administer sustained release (SR) bupropion 4 hours prior to receiving ECT. The investigators plan to compare the seizure threshold and seizure durations between ECT sessions with and without bupropion administration. The study's implication is to examine how ECT can be optimized by rational combination with medications that lower seizure threshold.

DETAILED DESCRIPTION:
Background and significance Depression is the leading cause of disability in individuals aged 15-44, resulting in 400 million disability days in a year (1). The total economic burden of the disease is estimated to be composed of $26.1 billion in direct medical costs, $5.4 billion in suicide-related mortality costs, and $51.5 billion in indirect workplace cost (1). Electroconvulsive therapy (ECT) is the gold-standard treatment for major depressive disorder (MDD) that is severe (2-5). The standard method of ECT used in the US now is right unilateral ultra-brief study. RUL ECT uses a pulse width of </= 0.3 ms, this optimizes electrical dosing and causes decreased severity of cognitive side effects. With right unilateral ECT it is essential for the stimulus to be above seizure threshold. The stimulus dosing is titrated to establish what seizure threshold is and this is titrated over the course of ECT sessions (6). Because the maximum ECT output is limited by FDA, a frequent problem encountered by ECT clinicians is high seizure threshold which at times cannot be provided by the ECT device and this compromises efficacy (7). Hence it would be useful to develop means to lower seizure threshold.

In addition, some studies show a reduction in efficacy with ultra-brief as compared to brief ECT with the former requiring higher number of ECTs to achieve remission in depression symptoms (8). There represents a need for increasing the efficacy for RUL ultra brief ECT given its favorable cognitive-side effect profile. Combining RUL ultra brief ECT with appropriate psychopharmacological agents to alter seizure profile is a feasible way of optimizing the efficacy.

Design and Procedures The study is designed to evaluate the effect of bupropion on seizure threshold in patients with major depressive disorder (MDD) referred for RUL ultra brief ECT. The study is powered to determine changes in seizure duration and seizure threshold by enrolling 10 subjects. The investigators plan to screen 20 subjects to have 10 participants. Potential participants will be discussed with the ECT team to which the patient would have been referred. Once a potential participant has been identified, a study team person will discuss the study and desire for participation in person with that individual during the ECT consult session which is needed prior to scheduling of the ECT session. If participants are found to be eligible they will be invited to participate in the study and the study will be initiated in conjunction with their first ECT session. Participants will go through the informed consent procedure. After providing informed consent participants will undergo a clinical assessment to confirm the inclusion/exclusion criteria.

Patients will receive ECT treatment as usual, but for this study if they choose to participate they will be randomized to receive bupropion (sustained release preparation 300 mg) (Wellbutrin ®), to be taken by mouth, in the morning (4 hours prior to ECT) on the day of ECT session 1 or session 2. There will be a one-time administration of bupropion at this dose with no discontinuation of medications that patient is already on. There will also be no washout period before bupropion administration or ECT.

The study is powered to determine changes in seizure duration and seizure threshold by enrolling 10 subjects (5 subjects will receive bupropion prior to ECT session 1 and 5 will receive it prior to ECT session 2). Counterbalanced randomization will be used to assign subject drug administration to ECT session 1 or 2 with inter-individual cross-over. The PI (Steven T Szabo Jr MD PhD) and coordinator (Gopalkumar Rakesh) would be blind to randomization details. Computer generated randomization would be done by Richard Weiner MD PhD - the director of the ECT program.

ECT administration The clinical procedure of ultra brief RUL ECT in these subjects will not be deviated from the usual procedure that is described below. ECT treatments will be provided three times a week, with standard right unilateral electrode placement with a MECTA spectrum device (MECTA Corporation, Portland, Ore.) with a pulse width </= 0.3 and a current of 0.8 A. A standard dose titration procedure to determine seizure threshold will be conducted at the first and second treatments, subjects would receive bupropion during one of these sessions. Subsequent treatments would be administered at 5.5 times seizure threshold from the treatment session without bupropion administration.

Clinical assessments The Montgomery-Asberg Depression Rating Scale (MADRS) is an assessment tool for depression symptom severity and will be carried out at baseline at every ECT visit. This is usual practice that the ECT clinician employs prior to the clinical administration of ECT. The investigators will also measure time to orientation recovery post ECT after the first and second ECT treatments.

Blood Collection During ECT sessions 1 and 2, just prior to administration of right unilateral (RUL) ECT, patients will be placed with a venous catheter and the investigators will acquire from consenting study patients a serum sample to be used to ascertain serum bupropion level.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, age >18.
2. Meeting diagnostic criteria for major depressive disorder or bipolar disorder per DSM5.
3. Referred for ultra brief RUL ECT.
4. Right motor dominant.
5. Competent to provide informed consent.
6. Able to read or comprehend English.
7. H/O treatment with bupropion.
8. Concomitant treatment with benzodiazepines, dosing of which has remained stable for a week prior to study ECT session.

Exclusion Criteria:

1. Lifetime history of schizophrenia, schizoaffective disorder, mental retardation, seizure disorder.
2. Current alcohol abuse or dependence within past 6 months.
3. Current substance abuse or dependence within past 6 months.
4. Recently received ECT within preceding 3-6 months.
5. Currently on any formulation of bupropion.
6. Currently on any anticonvulsants or clozapine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Szabo, MD PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenberg PE, Fournier AA, Sisitsky T, Pike CT, Kessler RC. The economic burden of adults with major depressive disorder in the United States (2005 and 2010). J Clin Psychiatry. 2015 Feb;76(2):155-62. doi: 10.4088/JCP.14m09298. PMID 25742202
- [Background] Beckford-Ball J. An overview of the new NICE guidelines on bipolar disorder. Nurs Times. 2006 Aug 22-28;102(34):23-4. PMID 16956074
- [Background] Fountoulakis KN, Vieta E, Sanchez-Moreno J, Kaprinis SG, Goikolea JM, Kaprinis GS. Treatment guidelines for bipolar disorder: a critical review. J Affect Disord. 2005 May;86(1):1-10. doi: 10.1016/j.jad.2005.01.004. PMID 15820265
- [Background] Frances AJ, Kahn DA, Carpenter D, Docherty JP, Donovan SL. The Expert Consensus Guidelines for treating depression in bipolar disorder. J Clin Psychiatry. 1998;59 Suppl 4:73-9. PMID 9554324
- [Background] Yatham LN, Kennedy SH, Parikh SV, Schaffer A, Beaulieu S, Alda M, O'Donovan C, Macqueen G, McIntyre RS, Sharma V, Ravindran A, Young LT, Milev R, Bond DJ, Frey BN, Goldstein BI, Lafer B, Birmaher B, Ha K, Nolen WA, Berk M. Canadian Network for Mood and Anxiety Treatments (CANMAT) and International Society for Bipolar Disorders (ISBD) collaborative update of CANMAT guidelines for the management of patients with bipolar disorder: update 2013. Bipolar Disord. 2013 Feb;15(1):1-44. doi: 10.1111/bdi.12025. Epub 2012 Dec 12. PMID 23237061
- [Background] Sackeim HA, Devanand DP, Prudic J. Stimulus intensity, seizure threshold, and seizure duration: impact on the efficacy and safety of electroconvulsive therapy. Psychiatr Clin North Am. 1991 Dec;14(4):803-43. PMID 1771150
- [Background] Lisanby SH, Devanand DP, Nobler MS, Prudic J, Mullen L, Sackeim HA. Exceptionally high seizure threshold: ECT device limitations. Convuls Ther. 1996 Sep;12(3):156-64. PMID 8872404
- [Background] Tor PC, Bautovich A, Wang MJ, Martin D, Harvey SB, Loo C. A Systematic Review and Meta-Analysis of Brief Versus Ultrabrief Right Unilateral Electroconvulsive Therapy for Depression. J Clin Psychiatry. 2015 Sep;76(9):e1092-8. doi: 10.4088/JCP.14r09145. PMID 26213985

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wellbutrin During ECT 1 | Wellbutrin During ECT 2
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wellbutrin During ECT 1 | Wellbutrin During ECT 2 | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (17.1) | 45.2 (6.5) | 47.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Seizure Threshold
Description: Charge in Millicoulombs at which subject gets a seizure with ECT. First measurement on day 1 of electroconvulsive treatment (ECT) and second measurement on day 2 of electroconvulsive therapy (ECT), separated by 1 day interval. This outcome measure was not measured at baseline.
Time Frame: Measured at day 1 and day 2
Measure: Mean (Standard Deviation); unit: millicoulombs
Arm/Group | Wellbutrin During ECT 1 | Wellbutrin During ECT 2
Number analyzed (Participants) | 5 | 5
millicoulombs | 23.04 (5.3) | 19.68 (6)

2. Primary Outcome: Change in Seizure Duration
Description: Duration of seizures with ECT. First measurement on day 1 of electroconvulsive treatment (ECT) and second measurement on day 2 of electroconvulsive therapy (ECT), separated by 1 day interval. This outcome measure was not measured at baseline.
Time Frame: Measured at day 1 and day 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Wellbutrin During ECT 1 | Wellbutrin During ECT 2
Number analyzed (Participants) | 5 | 5
seconds | 26.2 (14.1) | 29.6 (19.3)

3. Secondary Outcome: Change in MADRS Score
Description: Scoring of depressive symptoms on the Montgomery Asberg Depression Rating Scale, maximum 60 , minimum 0. Higher scores mean worse outcome. First measurement on day 1 of electroconvulsive treatment (ECT) and second measurement on day 2 of electroconvulsive therapy (ECT), separated by 1 day interval. This outcome measure was not measured at baseline.
Time Frame: Scored on day 1 and day 2 after ECT session
Measure: Mean (Standard Deviation); unit: Scored on a scale
Arm/Group | Wellbutrin During ECT 1 | Wellbutrin During ECT 2
Number analyzed (Participants) | 5 | 5
Scored on a scale | 2.60 (3.2) | 3.60 (3.4)
Statistical Analysis 1: Comparison: Wellbutrin During ECT 1 vs Wellbutrin During ECT 2; Test type: Superiority; p = 0.212, t-test, 2 sided — Threshold of <0.05

ADVERSE EVENTS:
Time Frame: Adverse events were assessed on days 1 and 2 of treatment and for a week after treatment 2.
Arm/Group | Wellbutrin During ECT 1 | Wellbutrin During ECT 2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT03126682/Prot_SAP_000.pdf